CLINICAL TRIAL: NCT04340973
Title: Comparing Different Transcranial Direct Current Stimulation Montages in Acute Stroke Patients: a Randomized, Triple-blinded, Sham-controlled Study
Brief Title: Comparing Transcranial Direct Current Stimulation Montages in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Assistant Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-94
Record Dates: First submitted 2020-04-04; First posted 2020-04-10 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Acute Stroke
Keywords: tDCS; Acute Stroke; WMFT; SWMT; Fugl Meyer
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 5 groups, each group receives one of four treatments or the sham treatment. Double-blinded, sham controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Everyone is blinded, codes are selected by a third party not involved in any step of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Anodal (Active Comparator): Anodal tDCS: Anode placer over the affected primary motor cortex, cathode over contralateral supra orbital area. 2 mA, 20min stimulation, 5 days a week for 4 weeks
  Interventions: Device: Transcranial Direct Current Stimulation
- Bilateral (Active Comparator): Bilateral : Anode placer over the affected primary motor cortex, cathode over unaffected motor cortex. 2 mA, 20min stimulation, 5 days a week for 4 weeks
  Interventions: Device: Transcranial Direct Current Stimulation
- Cathodal (Active Comparator): Cathodal : Cathode placer over the unaffected primary motor cortex, anode over contralateral supra orbital area. 2 mA, 20min stimulation, 5 days a week for 4 weeks
  Interventions: Device: Transcranial Direct Current Stimulation
- Extracephalic (Active Comparator): Extracephalic : Anode placer over the affected primary motor cortex, cathode over right shoulder. 2 mA, 20min stimulation, 5 days a week for 4 weeks
  Interventions: Device: Transcranial Direct Current Stimulation
- Placebo (Placebo Comparator): Placebo : anode montage but current is ramped up over 15 secondes, then ramped down. 2 mA, 20min stimulation, 5 days a week for 4 weeks
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Subjects received a micro-current through their scalp to induce cortical and subcortical changes
  Other Names: tDCS

SUMMARY:
40 acute subjects will be split into 5 groups. Each group will receive one of the following tDCS montages : anodal, bilateral, cathodal, extracephalic or placebo.

Subjects will receive, in addition to conventional rehabilitation, 2mA for 20 mins of their attributed tDCS, 5 times a week.

Evaluations will take place before the first stimulation period (48h post stroke), after 1, 2, 3 and 4 weeks. Evaluations consist of the Wolf Motor Function Test, the Fugl Meyer, and the Semmes Weinstein Monofilament Test

DETAILED DESCRIPTION:
40 acute subjects will be randomized and split into 5 groups.

Each group will receive one of the following tDCS montages :

Anodal : Anode placer over the affected primary motor cortex, cathode over contralateral supra orbital area Bilateral : Anode placer over the affected primary motor cortex, cathode over unaffected motor cortex Cathodal : Cathode placer over the unaffected primary motor cortex, anode over contralateral supra orbital area Extracephalic : Anode placer over the affected primary motor cortex, cathode over right shoulder Placebo : anode montage but current is ramped up over 15 secondes, then ramped down.

Subjects will receive, in addition to conventional rehabilitation (±1.5h/weekday), 2mA for 20 mins of their attributed tDCS, 5 times a week.

Evaluations will take place before the first stimulation period (48h post stroke), after 1, 2, 3 and 4 weeks. Evaluations consist of the Wolf Motor Function Test, the Fugl Meyer, and the Semmes Weinstein Monofilament Test

All researchers, therapists, data analysis and patients are blinded by a code system implemented in the tDCS machine

ELIGIBILITY:
Inclusion Criteria:

* First Ever Stroke
* Motor or sensory deficit
* Understands and follows orders
* Signed inform consent

Exclusion Criteria:

* One Yes on the medium and high risk sections of the TSST (Bornheim et al.,2019)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Wolf Motor Function Test | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  Functional upper limb test, filmed and scored subjectively
Change in Fugl Meyer Motor Assessment | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  Functional upper limb, lower limb and sensory test
Change in Semmes Weinstein Monofilament Test | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  11 Point Sensory test

CONTACTS AND LOCATIONS:
Locations (1):
- Liege Univeristy Hospital, Liège, Belgium

REFERENCES:
- [Background] Bornheim S, Croisier JL, Maquet P, Kaux JF. Proposal of a New Transcranial Direct Current Stimulation Safety Screening Tool. Am J Phys Med Rehabil. 2019 Jul;98(7):e77-e78. doi: 10.1097/PHM.0000000000001096. No abstract available. PMID 30431445